CLINICAL TRIAL: NCT00511095
Title: An Open-Label Study of Safety and Immunogenicity in Subjects Following Injection With Two Doses of HEPLISAV™
Brief Title: Open-Label Study of the Safety and Immunogenicity of HEPLISAV™ Hepatitis B Virus Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DV2-HBV-14
Record Dates: First submitted 2007-07-25; First posted 2007-08-03 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Hepatitis B
Keywords: Hepatitis B vaccine; HBV vaccine; Hepatitis B; Hepatitis; HBV; Vaccine; 1018; HBsAg
MeSH Terms: conditions — Hepatitis B; Hepatitis | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HEPLISAV (Experimental): 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018) Intramuscular (IM) injection 0.5mL
  Interventions: Biological: HEPLISAV

INTERVENTIONS:
Biological: HEPLISAV — Intramuscular (IM) injections 0.5mL on Day 0 and Week 4

SUMMARY:
The purpose of this study is to further evaluate the safety and seroprotective immune response of a new investigational hepatitis B virus (HBV) vaccine, HEPLISAV™, in subjects 11-55 years old. The primary hypothesis is that HEPLISAV™ is well tolerated.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of two injections of HEPLISAV™ in subjects 11 to 55 years old. About 200 subjects will be included in the study. Once subjects have been consented and screened, they will receive a total of two injections over a 28-day period, with follow-up visits at 8, 12 and 28 weeks. Safety and tolerability will be evaluated by occurrence of adverse events, periodic laboratory tests, vital signs, and local/systemic reactogenicity.

Comparison: This study does not include a control treatment; all subjects will receive treatment with HEPLISAV™.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Women of childbearing potential must be willing to consistently use a highly effective method of birth control

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Any previous HBV infection
* Previous vaccination (1 or more doses) with any HBV vaccine
* Any previous autoimmune diseases
* Are at high risk for recent exposure to HBV, Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV)
* Received any blood products or antibodies within 3 months prior to study entry
* Ever received an injection with DNA plasmids or oligonucleotides
* Received any vaccines within 4 weeks prior to study entry
* Received any other investigational medicinal agent within 4 weeks prior to study entry

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 207 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martins, MD, DPhil, Study Director — Dynavax Technologies Corporation
Locations (7):
- United States (7):
  - Beeghley Medical Park, Boardman, Ohio
  - Family Healthcare Partners, Grove City, Pennsylvania
  - Pediatric Alliance Southwestern, Pittsburgh, Pennsylvania
  - Primary Physicians Research, Pittsburgh, Pennsylvania
  - Family Practice Medical Associates South, Upper Saint Clair, Pennsylvania
  - The Washington Hospital Family Medicine, Washington, Pennsylvania
  - Metropolitan Research, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Dynavax Webpage — http://www.dynavax.com

RESULTS

PARTICIPANT FLOW:
Groups:
- HEPLISAV: 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018) HEPLISAV: Intramuscular (IM) injections at Week 0 and Week 4
Period: Overall Study
Arm/Group | HEPLISAV
Started | 207
Completed | 196
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | HEPLISAV
Number analyzed (Participants) | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 207
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133
  Male | 74
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 207

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local and Systemic Post-injection Reaction Rates
Description: Local and Systemic post-injection reactions.
Time Frame: Within 7 days post-injection for post-injection reactions at Week 0 and Week 4
Population: Safety Population: Subjects who received at least 1 study injection and had any post-baseline safety data
Measure: Number; unit: percentage of subjects
Groups:
- HEPLISAV (Week 0): 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018) HEPLISAV: Intramuscular (IM) injections at Week 0
- HEPLISAV (Week 4): 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018) HEPLISAV: Intramuscular (IM) injections at Week 4
Arm/Group | HEPLISAV (Week 0) | HEPLISAV (Week 4)
Number analyzed (Participants) | 207 | 203
percentage of subjects
  Local Reaction: Injection | 38.2 | 37.9
  Systemic Reaction: Injection | 37.2 | 33.0

2. Secondary Outcome: Percentage of Subjects Who Have a Seroprotective Immune Response (Anti-HBsAg ≥ 10 Milli-international Unit (mIU)/mL) at Weeks 4, 8, 12 and 28.
Description: Seroprotective Immune Response
Time Frame: Weeks 4, 8, 12 and 28
Population: Intent-to-treat population: Enrolled subjects who received at least 1 study injection irrespective of available immune response data.
Measure: Number; unit: percentage of subjects
Groups:
- HEPLISAV (Week 8): 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018) HEPLISAV: Intramuscular (IM) injections at Week 8
- HEPLISAV (Week 12): 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018) HEPLISAV: Intramuscular (IM) injections at Week 12
- HEPLISAV (Week 28): 0.5 mL HEPLISAV (20 mcg HBsAg and 3000 mcg 1018) HEPLISAV: Intramuscular (IM) injections at Week 28
Arm/Group | HEPLISAV (Week 4) | HEPLISAV (Week 8) | HEPLISAV (Week 12) | HEPLISAV (Week 28)
Number analyzed (Participants) | 205 | 199 | 198 | 196
percentage of subjects | 32.7 | 84.9 | 93.4 | 95.4

3. Secondary Outcome: Serum GMC of Anti-HBsAg Measured at Weeks 4, 8, 12, and 28
Description: Measurement of Serum GMC
Time Frame: Weeks 4, 8, 12, and 28
Population: Intent-to-treat population: Enrolled subjects who received at least 1 study injection irrespective of available immune response data.
  Note: "Number Analyzed" is the number of subjects with nonmissing concentrations at that visit.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HEPLISAV
Number analyzed (Participants) | 207
mIU/mL
  Week 4: number analyzed (Participants) | 205
  Week 4 | 11.5 [7.8 to 16.8]
  Week 8: number analyzed (Participants) | 199
  Week 8 | 97.1 [69.1 to 136.6]
  Week 12: number analyzed (Participants) | 198
  Week 12 | 170.7 [127.9 to 227.7]
  Week 28: number analyzed (Participants) | 196
  Week 28 | 349.4 [271.8 to 449.3]

ADVERSE EVENTS:
Arm/Group | HEPLISAV
Serious Adverse Events (participants affected / at risk) | 2/207
Other Adverse Events (participants affected / at risk) | 59/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV (N=207)
Hernia obstructive (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV (N=207)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 12
Headache (Nervous system disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less